CLINICAL TRIAL: NCT06767670
Title: Evaluation of Oral Hygiene Status in Correlation With Microbial Load in the Oral Cavity Following Restorations of Primary Molars Using Stainless Steel and Bioflex Crowns (Clinical Randomized Trial)
Brief Title: The Relation Between Oral Hygiene and Microbial Load in the Oral Cavity After Restoring Primary Molars With Two Types of Ready-made Crowns
Acronym: bioflex crown
Status: Recruiting | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Alaa M Eldehna, assistant proffesor, Al-Azhar University
Other Study IDs: P-PD-25-01
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Carious Lesion; Ready-made Crowns
Keywords: primary crowns,; oral health
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group S: teeth subjected to SSC on one side
  Interventions: Other: stainless steel crown
- Group B: teeth subjected to Bioflx crowns on the contralateral side
  Interventions: Other: bioflex crown

INTERVENTIONS:
Other: stainless steel crown — familiar method of managing multi-surface carious lesions in primary teeth
  Groups: Group S
Other: bioflex crown — aesthetic preformed pediatric crowns that offer the properties of both stainless steel and zirconia crowns
  Groups: Group B

SUMMARY:
Following the restoration of primary molars with stainless steel and bioflex crowns, an evaluation of the current state of oral hygiene in relation to the amount of microorganisms and gingival health in the oral cavity will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 4 and 8 years.
* Pulp therapy treated primary molars on the contralateral side, requiring a full coverage restoration (split-mouth technique).
* No history of any antibiotic consumption 2 weeks before the procedure.
* No history of fluoride application 2 weeks before the procedure.

Exclusion Criteria:

* Special children with physical disabilities or emotional disturbances.
* Children are diagnosed with systemic diseases.
* Grossly destructed teeth with non-restorable crown structure.
* Primary teeth with shedding or pathological tooth mobility.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A total of 10 patients 4-8 years old will be selected according to the established inclusion and exclusion criteria. The study will be conducted on patients attending the outpatient clinic of the pediatric dentistry department, Faculty of Dental Medicine Al-Azhar.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-06-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The adhesion of S. mutans to prefabricated Bioflx and Stainless-steel crowns under clinical conditions. | one months
  Collecting the plaque samples from the gingival crevices, buccal mucosa, and occlusal surfaces of the teeth treated using sterile cotton swabs initially and from the respective crown surfaces. After collecting the samples, they will be inoculated onto a plate of Mitis salivarius-bacitracin agar (MSBA), a selective growth medium for cultivating S. mutans.

SECONDARY OUTCOMES:
Gingival health | one months
  by measuring the gingival index (GI) Gingival Index (GI)
  * Purpose: Measures the severity of gingivitis based on the color, consistency, and bleeding of the gums.
  * Scoring:
    0: Normal gingiva
    1. Mild inflammation (slight change in color, slight edema, no bleeding).
    2. Moderate inflammation (redness, edema, and bleeding upon probing).
    3. Severe inflammation (marked redness and edema, spontaneous bleeding).
Plaque Index (PI) | one month
  * Purpose: Assesses the amount of dental plaque on teeth.
  * Scoring:
  No plaque
  1. A film of plaque adhering to the free gingival margin and adjacent areas of the tooth.
  2. Moderate accumulation of soft deposits on the gingival margin and/or the adjacent tooth surfaces.
  3. Abundance of soft matter on the tooth and gingival margin.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Mohammed Eldehna, Assistant Proffessor, Principal Investigator — Al-Azhar University
Locations (2):
- Egypt (2):
  - Al-Azhar University, Cairo, Nasr City
  - Faculty of Dental Medicine at Al-Azhar University., Cairo, Nasr City

IPD SHARING:
Plan to Share IPD: Undecided